CLINICAL TRIAL: NCT00576225
Title: Paclitaxel Poliglumex (CT-2103)/Carboplatin vs Paclitaxel/Carboplatin for the Treatment of Chemotherapy-Naïve Advanced Non-Small Cell Lung Cancer (NSCLC) in Women With Estradiol > 25 pg/mL
Brief Title: CT-2103/Carboplatin vs Paclitaxel/Carboplatin for NSCLC in Women With Estradiol > 25 pg/mL
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGT307
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: NSCLC
Keywords: NSCLC; women; CT-2103; paclitaxel; carboplatin
MeSH Terms: interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: CT-2103/carboplatin
- Control (Active Comparator)
  Interventions: Drug: paclitaxel/carboplatin

INTERVENTIONS:
Drug: CT-2103/carboplatin — CT-2103 (175 mg/m2 10 min IV infusion) and carboplatin (AUC 6, 30 min IV infusion) on day 1 of each 21-day cycle for up to 6 cycles.
  Arms: Experimental
Drug: paclitaxel/carboplatin — Paclitaxel (175 mg/m2, 3 hr IV infusion) and carboplatin (AUC 6) (30 minute IV infusion) on day 1 of each 21-day cycle for up to 6 cycles.
  Arms: Control

SUMMARY:
This study is designed to test whether CT-2103/carboplatin provides improved overall survival compared to paclitaxel/carboplatin in women with NSCLC who have estradiol levels >30 pg/ml.

ELIGIBILITY:
Inclusion Criteria:

1. Women with baseline estradiol >25 pg/mL
2. Histologically- or cytologically-confirmed diagnosis of NSCLC.
3. ECOG performance score (PS) of 0, 1, or 2.
4. Patients must meet one of the following criteria have either (1) Recurrent disease following completion of radiation or surgery, (2) Stage IIIB disease and not be a candidate for combined modality therapy (primary radiation therapy or surgery), or (3) Stage IV disease.
5. At least 18 years of age.
6. Adequate bone marrow function
7. Adequate renal function
8. Adequate hepatic function
9. Life expectancy ≥12 weeks

Exclusion Criteria:

1. Known hypersensitivity to the excipients or the study drug (either CT-2103, paclitaxel, or carboplatin that the patient will receive.
2. Evidence of small cell carcinoma, carcinoid, or mixed small cell/non-small cell histology.
3. Weight loss >10% in previous 6 months
4. LDH > 2.5X IULN
5. Both LDH > 1.5X IULN and ≥ 5% weight loss in previous 6 months
6. BMI >35
7. Any prior systemic chemotherapy for the treatment of lung cancer. This includes systemic radiosensitizers used to treat brain metastases and any biologic agent.
8. Local palliative radiotherapy < 7 days before randomization.
9. Radiation with curative intent < 30 days before randomization.
10. Concurrent primary malignancies except for carcinoma in situ or non-melanoma skin cancer.
11. Grade 2 or greater neuropathy.
12. Evidence of significant unstable neurological symptoms within the 4 weeks before study randomization.
13. Clinically significant active infection for which active therapy is underway.
14. Investigational therapy within 4 weeks before randomization, unless local requirements are more stringent.
15. Unstable medical conditions including unstable angina or myocardial infarction within the past 6 months before randomization.
16. Pregnant women or nursing mothers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2010-04-05 (Actual); Study Completion 2010-04-05 (Actual)

PRIMARY OUTCOMES:
Survival | up to 3 years post treatment

SECONDARY OUTCOMES:
progression-free survival, disease control, clinical benefit, response rate, quality of life, and the safety | up to 3 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jack W. Singer, M.D., Study Director — CTI BioPharma
Locations (44):
- United States (44):
  - Scottsdale Medical Specialists, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Hembree Regional Cancer Center, Fort Smith, Arkansas
  - Providence St. Joseph Medical Center, Burbank, California
  - Southwest Cancer Care, Escondido, California
  - Clinical Trials & Research Institute, Montebello, California
  - Stanford Cancer Center, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Horizon Institute for Clinical Research, Hollywood, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Pasco Pinellas Cancer Center, Tarpon Springs, Florida
  - Joliet Oncology Hematology Associates, Ltd, Joliet, Illinois
  - Loyola University, Maywood, Illinois
  - Hematology Oncology Consultants, Naperville, Illinois
  - Cancer Care Center, New Albany, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Family Medicine of Vincennes Clinical Trials Center, Vincennes, Indiana
  - Kansas City Cancer Center, Overland Park, Kansas
  - Henry Ford Health System, Josephine Ford Cancer Center, Detroit, Michigan
  - W. Michigan Regional Cancer & Blood Center, Free Soil, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Columbia Comprehensive Cancer Care Clinics, Jefferson City, Missouri
  - St. Louis University, St Louis, Missouri
  - Las Vegas Cancer Center, Henderson, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Lincoln Medical and Mental Health Center, New York, New York
  - Arena Oncology Associates, New York, New York
  - Richmond University Medical Center, Staten Island, New York
  - New York Medical College, Valhalla, New York
  - St Alexius Medical Center, Bismarck, North Dakota
  - Blood and Cancer Center, Canfield, Ohio
  - Aultman Hospital Clinical Trials, Canton, Ohio
  - UIMA, Inc / University of Cincinnati-Barrett Cancer Center, Cincinnati, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Vita Hematology Oncology, P.C., Fountain Hill, Pennsylvania
  - The Family Cancer Center, Collierville, Tennessee
  - Mid-South Cancer Center, Germantown, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - Lone Star Oncology Consultants, Austin, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Northern Utah Associates, Ogden, Utah
  - Cancer Outreach Associates, LLC, Arlington, Virginia
  - Virginia Mason Medical Center, Seattle, Washington